CLINICAL TRIAL: NCT03758638
Title: Disseminating and Implementing A Lifestyle Based Healthy Weight Program in a National Organization
Brief Title: Healthy Eating and Active Living Taught at Home (HEALTH) Dissemination & Implementation (D&I)
Acronym: HEALTH D&I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 201810157-1R01HL143360
Record Dates: First submitted 2018-11-26; First posted 2018-11-29 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Diet, Healthy

STUDY DESIGN:
Intervention Model Description: Healthy Eating & Active Living Taught at Home (HEALTH) embeds content related to healthy eating and activity within Parents as Teachers (PAT)'s existing home visits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Eating & Active Living Taught at Home (Experimental): PAT National Center will train educators affiliated with PAT sites in HEALTH; among these, using the HEALTH training curriculum (implementation strategy).
  Participants at HEALTH sites receive usual care PAT+evidence-based life-style change strategies to prevent weight gain and promote weight loss embedded within and delivered as part of home visits.
  Interventions: Behavioral: Healthy Eating & Active Living Taught at Home
- Usual Care (Active Comparator): Participants at usual care PAT sites will receive PAT as usual
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: Healthy Eating & Active Living Taught at Home — PAT National Center will train educators affiliated with PAT sites in HEALTH; among these, using the HEALTH training curriculum, which includes training materials, an ~8 hour training delivered through a synchronous web-based experience, and ongoing consultation. Participants at HEALTH sites receive usual care PAT+evidence-based life-style change strategies to prevent weight gain and promote weight loss embedded within and delivered as part of home visits. In addition to the usual care PAT curriculum content, goal setting related to healthy weight, and the importance of parental modeling of healthy eating and physical activity are incorporated throughout the discussion and visit. HEALTH will be delivered over 24 months via a (1) core and (2) maintenance phase. The visits begin with greater frequency, and taper. Consistent with PAT practice, the frequency and number of visits are determined by the family's needs and preferences.
  Arms: Healthy Eating & Active Living Taught at Home
Behavioral: Usual Care — The Foundational (usual care) curriculum uses a strength-based, solution-focused model to provide parents with child development knowledge and parenting support, empowering parents as their child's first and most influential teacher.
  Other Names: Parents as Teachers
  Arms: Usual Care

SUMMARY:
This project evaluates the effectiveness of an evidence-based intervention (HEALTH) to prevent weight gain and promote weight loss when disseminated and implemented in real-world settings, through Parents as Teachers. To enhance the impact of HEALTH, the study also evaluates implementation outcomes from the training curriculum (implementation strategy) and external validity when HEALTH is implemented within this national home visiting organization. This partnership has potential for significant impact on obesity and chronic diseases such as cardiovascular disease and diabetes.

DETAILED DESCRIPTION:
Excessive weight gain among young adult women age 18-35 years is an alarming and overlooked trend that must be addressed to reverse the epidemics of obesity and chronic disease. During this vulnerable period women tend to gain disproportionally large amounts of weight compared to men and other life periods. A lifestyle modification intervention (HEALTH) that prevented weight gain, promoted sustained weight loss, and reduced waist circumference was developed in partnership with Parents as Teachers (PAT), a national home visiting, community based organization with significant reach in this population. PAT provides parent-child education and services free-of-charge to nearly 170,000 families through up to 25 free home visits per year until the child enters kindergarten. This study will extend these findings with a pragmatic cluster randomized controlled trial to evaluate dissemination and implementation of HEALTH across three levels (mother, parent educator, PAT site) to achieve widespread impact. The pragmatic cluster randomized controlled trial will evaluate HEALTH and the HEALTH training curriculum (implementation strategy) on weight among mothers with overweight and obesity across the US (N= 200 HEALTH; N= 200 usual care). Parent educators from 40 existing PAT sites (20 HEALTH, 20 usual care) will receive the HEALTH training curriculum through the PAT National Center, using PAT's existing training infrastructure, as a continuing education opportunity. An extensive evaluation, guided by RE-AIM (Reach, Efficacy, Adoption, Implementation, and Maintenance) will determine implementation outcomes (acceptability, adoption, appropriateness, feasibility, fidelity, and adaptation) at the parent educator level. The Conceptual Framework for Implementation research will characterize determinants that influence HEALTH dissemination and implementation at three levels: mother, parent educator, PAT site to enhance external validity (reach and maintenance) and population level impact. The findings from this innovative study will have significant potential to help reverse the trend of excessive weight gain among young adult women, a critical priority target in battling the epidemics of obesity and chronic disease, by reaching women with an evidence-based intervention nation-wide.

ELIGIBILITY:
For Parent educators:

Inclusion Criteria:

* Deliver PAT at a site participating in the study
* Provide informed consent

Exclusion Criteria:

* At least 18 years of age

For Participants:

Inclusion Criteria:

* 18-45 years of age
* overweight or obese (BMI 25-45 kg/m2)
* English or Spanish speaking
* participating or willing to participate in PAT at a participating PAT site for 2 years
* able to give informed consent for participation

Exclusion Criteria:

* currently pregnant or planning to become pregnant in the next 24 months
* unable to speak English or Spanish
* unable to engage in a walking program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — For the participants (i.e., not the parent educators), only women will be included: Including only female participants is scientifically justified, as the study focus is addressing the dramatic weight gain women experience in early adulthood, which is not experienced to the same extent among men. Further, HEALTH was tested and demonstrated effectiveness only in mothers, and the very small number of fathers who participate in PAT will not provide an adequate sample to evaluate HEALTH in this population.
Enrollment: 620 (Actual)
Dates: Start 2019-01-25 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2025-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel G Tabak, PhD, RD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St. Louis, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided
* Only data with identifiers removed will be shared publicly.
  * Any identified data to be shared will only be done so in coordination with the Human Research Protection Office at Washington University in St. Louis and the Institutional Review Board (IRB) at the requesting investigator's institution.
  * Datasets with identifiers will only be accessible to study team members with appropriate Human Subjects training.

REFERENCES:
- [Derived] Gilbert A, Martinez A, Farabi S, Cortez A, Baumann AA, Haire-Joshu D, Brownson RC, Morshed AB, Tabak RG. Social determinants of health influence maternal health behaviors and engagement in an obesity prevention intervention. Transl Behav Med. 2026 Jan 7;16(1):ibaf088. doi: 10.1093/tbm/ibaf088. PMID 41498407
- [Derived] Tabak RG, Schwarz CD, Kemner A, Haire-Joshu D. Cross-Sectional associations between inner setting determinants of self-efficacy and intent to deliver a healthy eating and activity curriculum embedded in a community setting. Int J Behav Nutr Phys Act. 2025 Apr 10;22(1):42. doi: 10.1186/s12966-025-01736-5. PMID 40211363
- [Derived] Farabi SS, Schwarz C, Persaud A, Gilbert A, Haire-Joshu D, Tabak RG. Sleep, Stress, and Cardiometabolic Health in Women of Childbearing Age with Overweight and Obesity. Womens Health Rep (New Rochelle). 2024 Feb 21;5(1):143-151. doi: 10.1089/whr.2023.0138. eCollection 2024. PMID 38414886
- [Derived] Tabak RG, Schwarz CD, Kemner A, Johnston S, Aramburu A, Haire-Joshu D. Social Determinants of Health Discussed with Mothers During Personal Visits Before and During the COVID-19 Pandemic. Health Equity. 2021 Sep 3;5(1):536-544. doi: 10.1089/heq.2020.0140. eCollection 2021. PMID 34909520
- [Derived] Tabak RG, Schwarz CD, Kemner A, Schechtman KB, Steger-May K, Byrth V, Haire-Joshu D. Disseminating and implementing a lifestyle-based healthy weight program for mothers in a national organization: a study protocol for a cluster randomized trial. Implement Sci. 2019 Jun 25;14(1):68. doi: 10.1186/s13012-019-0916-0. PMID 31238955

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Eating & Active Living Taught at Home: PAT National Center will train educators affiliated with PAT sites in HEALTH; among these, using the HEALTH training curriculum (implementation strategy).
  Participants at HEALTH sites receive usual care PAT+evidence-based life-style change strategies to prevent weight gain and promote weight loss embedded within and delivered as part of home visits.
  Healthy Eating & Active Living Taught at Home: PAT National Center will train educators affiliated with PAT sites in HEALTH; among these, using the HEALTH training curriculum, which includes training materials, an ~8 hour training delivered through a synchronous web-based experience, and ongoing consultation. Participants at HEALTH sites receive usual care PAT+evidence-based life-style change strategies to prevent weight gain and promote weight loss embedded within and delivered as part of home visits. In addition to the usual care PAT curriculum content, goal setting related to healthy weight, and the importance of parental modeling of healthy eating and physical activity are incorporated throughout the discussion and visit. HEALTH will be delivered over 24 months via a (1) core and (2) maintenance phase. The visits begin with greater frequency, and taper. Consistent with PAT practice, the frequency and number of visits are determined by the family's needs and preferences.
Period: Overall Study
Arm/Group | Healthy Eating & Active Living Taught at Home | Usual Care
Started | 349 | 271
Completed | 79 | 62
Not Completed | 270 | 209
Not completed — Pregnancy | 17 | 25
Not completed — Lost to Follow-up | 60 | 54
Not completed — Protocol Violation | 2 | 0
Not completed — Withdrawal by Subject | 8 | 2
Not completed — Providers not included in the primary outcome. | 183 | 128

BASELINE CHARACTERISTICS:
Population: As a dissemination and implementation trial, the current study includes outcomes at the parent level (n=309) as well as the perspectives of the providers (n=311) delivering the intervention. Since these providers completed data collection (e.g., their perspectives of the intervention) these 311 individuals were considered human subjects and enrolled in the study. However, the focus of the primary outcome is on the weight outcomes among the 309 parents.
Groups:
- Total: Total of all reporting groups
Arm/Group | Healthy Eating & Active Living Taught at Home | Usual Care | Total
Number analyzed (Participants) | 349 | 271 | 620
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: As a dissemination and implementation trial, the current study includes outcomes at the parent level (n=309) as well as the perspectives of the providers (n=311) delivering the intervention. Since these providers completed data collection (e.g., their perspectives of the intervention) these 311 individuals were considered human subjects and enrolled in the study. However, the focus of the primary outcome is on the weight outcomes among the 309 parents.
  Years
    Age of participant: number analyzed (Participants) | 166 | 143 | 309
    Age of participant | 30.3 (5.6) | 31.2 (6.1) | 30.7 (5.8)
    Age of provider: number analyzed (Participants) | 183 | 128 | 311
    Age of provider | 39.75 (12.05) | 40.11 (12.04) | 39.93 (12.05)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: As a dissemination and implementation trial, the current study includes outcomes at the parent level (n=309) as well as the perspectives of the providers (n=311) delivering the intervention. Since these providers completed data collection (e.g., their perspectives of the intervention) these 311 individuals were considered human subjects and enrolled in the study. However, the focus of the primary outcome is on the weight outcomes among the 309 parents.
  Participants
    Sex of participant: number analyzed (Participants) | 166 | 143 | 309
    Sex of participant: Female | 166 | 143 | 309
    Sex of participant: Male | 0 | 0 | 0
    Sex of provider: number analyzed (Participants) | 183 | 128 | 311
    Sex of provider: Female | 182 | 128 | 310
    Sex of provider: Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: As a dissemination and implementation trial, the current study includes outcomes at the parent level (n=309) as well as the perspectives of the providers (n=311) delivering the intervention. Since these providers completed data collection (e.g., their perspectives of the intervention) these 311 individuals were considered human subjects and enrolled in the study. However, the focus of the primary outcome is on the weight outcomes among the 309 parents.
  Participants
    Ethnicity of participant: number analyzed (Participants) | 166 | 143 | 309
    Ethnicity of participant: Hispanic or Latino | 68 | 62 | 130
    Ethnicity of participant: Not Hispanic or Latino | 89 | 67 | 156
    Ethnicity of participant: Unknown or Not Reported | 9 | 14 | 23
    Ethnicity of provider: number analyzed (Participants) | 183 | 128 | 311
    Ethnicity of provider: Hispanic or Latino | 58 | 36 | 94
    Ethnicity of provider: Not Hispanic or Latino | 114 | 80 | 194
    Ethnicity of provider: Unknown or Not Reported | 11 | 12 | 23
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: As a dissemination and implementation trial, the current study includes outcomes at the parent level (n=309) as well as the perspectives of the providers (n=311) delivering the intervention. Since these providers completed data collection (e.g., their perspectives of the intervention) these 311 individuals were considered human subjects and enrolled in the study. However, the focus of the primary outcome is on the weight outcomes among the 309 parents.
  Participants
    Race of participants: number analyzed (Participants) | 166 | 143 | 309
    Race of participants: American Indian or Alaska Native | 0 | 1 | 1
    Race of participants: Asian | 4 | 1 | 5
    Race of participants: Native Hawaiian or Other Pacific Islander | 1 | 2 | 3
    Race of participants: Black or African American | 25 | 15 | 40
    Race of participants: White | 93 | 66 | 159
    Race of participants: More than one race | 5 | 9 | 14
    Race of participants: Unknown or Not Reported | 38 | 49 | 87
    Race of providers: number analyzed (Participants) | 183 | 128 | 311
    Race of providers: American Indian or Alaska Native | 0 | 0 | 0
    Race of providers: Asian | 1 | 2 | 3
    Race of providers: Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
    Race of providers: Black or African American | 20 | 10 | 30
    Race of providers: White | 128 | 88 | 216
    Race of providers: More than one race | 6 | 0 | 6
    Race of providers: Unknown or Not Reported | 26 | 28 | 54
Baseline Weight [Median (Inter-Quartile Range); unit: Kg] — Population: As a dissemination and implementation trial, the current study includes outcomes at the parent level (n=309) as well as the perspectives of the providers (n=311) delivering the intervention. Since these providers completed data collection (e.g., their perspectives of the intervention) these 311 individuals were considered human subjects and enrolled in the study. However, the focus of the primary outcome is on the weight outcomes among the 309 parents.
  Kg
    Weight of participants: number analyzed (Participants) | 166 | 143 | 309
    Weight of participants | 83.6 [73.6 to 97.5] | 79.7 [73.0 to 99.3] | 81.4 [73.1 to 98.4]
    Weight of providers: number analyzed (Participants) | 161 | 114 | 275
    Weight of providers | 78.02 [65.77 to 91.17] | 76.66 [63.50 to 95.25] | 77.11 [63.96 to 92.53]

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Mother's body weight assessed by data collector
Time Frame: 24-months
Measure: Mean (Standard Deviation); unit: Kg
Arm/Group | Healthy Eating & Active Living Taught at Home | Usual Care
Number analyzed (Participants) | 79 | 62
Kg | -0.24 (9.75) | 0.49 (11.87)

2. Secondary Outcome: Fidelity of Delivery to the Intervention
Description: Parent educators' fidelity to the intervention will all be assessed using a coding document (developed for the current study), which will be applied to audio-recordings of study visits, and will document the following components: adherence, quality of delivery, exposure to the intervention, and participant responsiveness or involvement, all of which share a common unit of measure
Time Frame: throughout intervention delivery, which can range from 2-4 years for parent educators depending on when their site is randomized
Measure: Count of Units; unit: Visit recordings
Units Other Than Participants: Visit recordings
Arm/Group | Healthy Eating & Active Living Taught at Home
Number analyzed (Participants) | 20
Number analyzed (Visit recordings) | 88
Visit recordings
  High | 67
  Low | 12
  Other/NA/Missing | 9

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Healthy Eating & Active Living Taught at Home | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/349 | 0/271
Serious Adverse Events (participants affected / at risk) | 0/349 | 0/271
Other Adverse Events (participants affected / at risk) | 0/349 | 0/271

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-17): https://cdn.clinicaltrials.gov/large-docs/38/NCT03758638/Prot_SAP_000.pdf
  • Informed Consent Form (2020-10-05): https://cdn.clinicaltrials.gov/large-docs/38/NCT03758638/ICF_001.pdf